CLINICAL TRIAL: NCT02260921
Title: A Multi-Center, Prospective, Double-Blind, Randomized Controlled Study to Evaluate the Effectiveness and Safety of the Iovera° Device for the Temporary Relief of Pain Associated With Knee Osteoarthritis
Brief Title: Study to Evaluate the Iovera° Device for Temporary Relief From Knee Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pacira Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MYO-0946
Record Dates: First submitted 2014-10-03; First posted 2014-10-09 (Estimated); Results first posted 2020-12-31 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- iovera° Treatment (Experimental): Treatment with the iovera° device administered by a trained investigator to treat knee pain.
  Interventions: Device: iovera°
- Sham Treatment (Sham Comparator): Sham Treatment (similar device with no active therapeutic treatment) administered by a trained investigator to treat knee pain.
  Interventions: Device: Sham Comparator

INTERVENTIONS:
Device: iovera°
  Arms: iovera° Treatment
Device: Sham Comparator
  Arms: Sham Treatment

SUMMARY:
This purpose of this study is to evaluate the effectiveness and safety of the iovera° device for the temporary reduction of pain associated with knee osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

* 35 - 75 years of age
* American College of Rheumatology (ACR) criteria for osteoarthritis of the knee. This includes radiographic evidence of osteophytes and at least one of the following: age ≥ 50 years old, morning stiffness ≤ 30 minute duration or crepitus on motion.
* Grade II or III osteoarthritis of the knee as determined by Kellgren-Lawrence classification grading scale on anteroposterior (AP) x-ray within previous 6 months.
* Participants are ambulatory without assistive devices.
* Knee pain of ≥ 40 mm on Visual Analog Scale (VAS) when performing one of two movements that elicit the worst pain: standing from a seated position or walking up/down stairs.
* Participant reports knee pain in the anterior and/or inferior aspect of the knee as documented on the knee pain map in the appropriate areas.
* A diagnostic lidocaine (without epinephrine) block of the infrapatellar branch of the saphenous nerve results in a 50% reduction in the VAS pain assessment score when performing the activity that elicits the worst pain: standing from a seated position or walking up/down stairs.
* Participant is able to tolerate a washout of prescription and over-the-counter pain relief for a duration of 5 times the half-life of the medication prior to the Baseline visit.

Participant is able to tolerate a washout of adjunctive therapies for knee pain for 72 hours prior to the Baseline visit.

* Western Ontario and McMaster Osteoarthritis Index (WOMAC) NRS3.1 Pain subscore ≥ 20 at Baseline/Visit 2.
* Participant is able to tolerate discontinuation of all pain medication throughout the duration of the study. Acetaminophen may be used as rescue medication with a maximum dose of 4g per day.
* Participant is able to tolerate discontinuation of rescue medication, acetaminophen, for 24 hours prior to all follow-up visits.
* Prescription and over-the-counter pain medications must be maintained on a stable schedule for at least two weeks prior to screening.
* Participant is willing and able to give written informed consent.
* Participant is willing and able to comply with study instructions and commit to all follow-up visits for the duration of the study.
* Participant is in good general health and free of any systemic disease state or physical condition that might impair evaluation or which in the Investigator's opinion, exposes the Participant to an unacceptable risk by study participation.

Exclusion Criteria:

* History of a partial or full knee replacement of the knee to be treated.
* Planned partial or full knee replacement within the next 12 months in knee to be treated.
* Previous myoscience Focused Cold Therapy^TM (FCTTM) treatment.
* Viscosupplementation within the previous 6 months in knee to be treated.
* Participant reports the majority of knee pain outside of the anterior/inferior aspect of the knee.
* Intra-articular steroid injection in the knee to be treated within previous 3 months.
* Gross deformity of the knee including varus or valgus.
* Started physical therapy of the knee to be treated within 3 months of screening.
* Received acupuncture for knee pain within 3 months prior to screening.
* Body Mass Index ≥ 35.
* Prior surgery in the treatment area that may alter the anatomy of the infrapatellar branch of the saphenous nerve or result in scar tissue in the treatment area.
* Open and/or infected wound in the treatment area.
* Disease of the spine, hip, contralateral knee or other lower extremity joint of sufficient degree affecting the assessment of the treated knee.
* Acetaminophen intolerance or allergy.
* Allergy to lidocaine.
* History of cryoglobulinemia
* History of paroxysmal cold hemoglobinuria.
* History of cold urticaria.
* History of Raynaud's disease.
* History of pes anserinus bursitis in the knee to be treated.
* Use of extended-release or long-acting opioids within previous 3 months.
* Use of immediate-release opioids for more than 3 days per week within previous month.
* Participant is pregnant or planning to become pregnant while enrolled in the study.
* Current enrollment in any investigational drug or device study or participation within 30 days prior to screening.
* Any additional diagnosis that in the opinion of the Investigator directly contributes to knee pain.
* Any concomitant inflammatory disease or other condition that affects the joints (e.g. rheumatoid arthritis, metabolic bone disease, gout, active infection, etc.)
* Any clotting disorder and/or use of an anticoagulant (e.g., aspirin, warfarin, clopidogrel, etc.) within seven (7) days prior to administration of the device.
* Any local skin condition at the treatment site that in the Investigator's opinion would adversely affect treatment or outcomes.
* Any chronic medical condition that in the Investigator's opinion would prevent adequate participation.
* Any chronic medication use (prescription, over-the-counter, etc.) that in the Investigator's opinion would affect study participation or Subject safety.
* For any reason, in the opinion of the Investigator, the Subject may not be a suitable candidate for study participation (i.e., history of noncompliance, drug dependency, any related knee injury due to a worker's compensation claim, etc.).
* Known liver dysfunction.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2014-10-20 (Actual); Primary Completion 2016-02 (Actual); Study Completion 2016-05-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (17):
- United States (17):
  - Medvin Clinical Research, Covina, California
  - UC Davis Center for Musculoskeletal Health, Sacramento, California
  - Coastal Orthopedics and Sports Medicine of Southwest Florida, PA, Bradenton, Florida
  - Shrock Orthpedic Research, Fort Lauderdale, Florida
  - Health Awareness, Jupiter, Florida
  - JM Clinical Research, South Miami, Florida
  - Injury Care Medical Center, Boise, Idaho
  - Rockford Orthopedic Associates, LTD, Rockford, Illinois
  - Kansas University Medical Center, Fairway, Kansas
  - Kansas City Bone and Joint Clinic, Overland Park, Kansas
  - Covington Orthopedic and Sports Medicine Institute, Covington, Louisiana
  - LHU HSC Department of Orthopaedics, New Orleans, Louisiana
  - Arthritis Treatment Center, Frederick, Maryland
  - Triangle Orthopaedic Associates, P.A., Durham, North Carolina
  - Blair Orthopedic Associates, Inc., Altoona, Pennsylvania
  - PCET Research Center, Knoxville, Tennessee
  - Spokane Joint Replacement Center, Spokane, Washington

REFERENCES:
- [Derived] Radnovich R, Scott D, Patel AT, Olson R, Dasa V, Segal N, Lane NE, Shrock K, Naranjo J, Darr K, Surowitz R, Choo J, Valadie A, Harrell R, Wei N, Metyas S. Cryoneurolysis to treat the pain and symptoms of knee osteoarthritis: a multicenter, randomized, double-blind, sham-controlled trial. Osteoarthritis Cartilage. 2017 Aug;25(8):1247-1256. doi: 10.1016/j.joca.2017.03.006. Epub 2017 Mar 20. PMID 28336454

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Iovera° Treatment | Sham Treatment
Started | 121 | 59
Per-Protocol Population | 112 | 56
Completed | 107 | 55
Not Completed | 14 | 4
Not completed — Adverse Event | 1 | 0
Not completed — Lost to Follow-up | 4 | 3
Not completed — Withdraw Consent | 4 | 1
Not completed — Death | 1 | 0
Not completed — Prohibited Treatment for Knee Pain | 4 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) Analysis Population include all randomized participants who underwent the assigned treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Iovera° Treatment | Sham Treatment | Total
Number analyzed (Participants) | 121 | 59 | 180
Age, Continuous [Mean (Full Range); unit: years] | 60.7 [36.5 to 75.3] | 61.3 [40.3 to 74.7] | 61.0 [36.5 to 75.3]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 79 | 40 | 119
  Male | 42 | 19 | 61
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 8 | 8 | 16
  White | 110 | 50 | 160
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 121 | 59 | 180
Body Mass Index (BMI) [Median (Full Range); unit: kg/m^2] | 29.02 [18.6 to 41.4] | 29.99 [20.3 to 35.5] | 29.5 [18.6 to 41.4]

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change From Baseline in Western Ontario and McMaster Universities Arthritis Index (WOMAC) Pain Subscale Score at Day 30
Description: The WOMAC is a tri-dimensional, disease-specific, patient-reported outcome measure. It consists of 24 questions [each question is presented in a numerical rating scale format with possible values between 0= No (best) to 10= Extreme (worst)] with 5 questions regarding pain [possible subscale score 0 to 50], 2 questions regarding stiffness [possible subscale score 0 to 20] and 17 questions regarding function difficulty [possible subscale score 0 to 170]. A negative change from Baseline indicates improvement. An Analysis of Covariance (ANCOVA) model was used for analyses.
Time Frame: Baseline to Day 30
Population: Per-protocol Analysis Population included all participants who were randomized and underwent the assigned treatment where the treatment was successfully delivered as intended by the device and who are compliant with wash-out of pain medication prior to Baseline visit prior to study visit analyzed.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Iovera° Treatment | Sham Treatment
Number analyzed (Participants) | 112 | 56
score on a scale | -16.33 (1.15) | -8.79 (1.63)
Statistical Analysis 1: Comparison: Iovera° Treatment vs Sham Treatment; Test type: Superiority; p = 0.0002, ANCOVA — P-values are obtained by fitting an ANCOVA model with treatment as factor and WOMAC baseline pain score as a covariate; Difference in Least Squares (LS) Means = -7.53, 95% CI 2-sided [-11.48 to -3.58] — LS estimates are obtained by fitting an ANCOVA model with treatment as factor and WOMAC baseline pain score as a covariate

2. Secondary Outcome: Change From Baseline in Visual Analog Scale (VAS) at Day 30
Description: VAS pain assessment is a measure of pain intensity. The scale is made up of a 10 centimeter (cm) [100 millimeter (mm)] horizontal line. The far left of the horizontal line is labeled "no pain" while the far right of the horizontal line is labeled "worst imaginable pain". A negative change from Baseline indicates improvement. An ANCOVA model was used for analyses.
Time Frame: Baseline to Day 30
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Iovera° Treatment | Sham Treatment
Number analyzed (Participants) | 112 | 56
score on a scale | -39.20 (2.74) | -25.70 (3.89)

3. Secondary Outcome: Change From Baseline in Total WOMAC Score at Day 30
Description: The WOMAC is a tri-dimensional, disease-specific, patient-reported outcome measure. It consists of 24 questions [each question is presented in a numerical rating scale format with possible values between 0= No (best) to 10= Extreme (worst)] with 5 questions regarding pain [possible subscale score 0 to 50], 2 questions regarding stiffness [possible subscale score 0 to 20] and 17 questions regarding function difficulty [possible subscale score 0 to 170]. The WOMAC total score was calculated by summing the 3 subscales for a total possible score of 0 to 240. A negative change from Baseline indicates improvement. An ANCOVA model was used for analyses.
Time Frame: Baseline to Day 30
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Iovera° Treatment | Sham Treatment
Number analyzed (Participants) | 112 | 56
score on a scale | -77.18 (5.38) | -43.77 (7.61)

4. Secondary Outcome: Change From Baseline in VAS at Day 60
Description: VAS pain assessment is a measure of pain intensity. The scale is made up of a 10 cm (100 mm) horizontal line. The far left of the horizontal line is labeled "no pain" while the far right of the horizontal line is labeled "worst imaginable pain". A negative change from Baseline indicates improvement. An ANCOVA model was used for analyses.
Time Frame: Baseline to Day 60
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Iovera° Treatment | Sham Treatment
Number analyzed (Participants) | 112 | 56
score on a scale | -37.46 (2.80) | -28.82 (3.97)

5. Secondary Outcome: WOMAC Pain Score Responder Rate at Day 30
Description: WOMAC Pain Score Responder Rate is defined as the percentage of participants with at least a 30% reduction in the WOMAC pain score at Day 30 compared to Baseline. WOMAC is a tri-dimensional, disease-specific, patient-reported outcome measure. It consists of 24 questions [each question is presented in a numerical rating scale format with possible values between 0= No to 10= Extreme] with the first 5 questions regarding pain [possible subscale score 0 (best) to 50 (worst)].
Time Frame: Day 30
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Iovera° Treatment | Sham Treatment
Number analyzed (Participants) | 112 | 56
percentage of participants | 67.9 | 44.6

6. Secondary Outcome: VAS Responder Rate at Day 30
Description: VAS Responder Rate is defined as the percentage of participants with at least a 30% reduction in VAS at Day 30 compared to Baseline VAS pain assessment is a measure of pain intensity. The scale is made up of a 10 cm (100 mm) horizontal line. The far left of the horizontal line is labeled "no pain" while the far right of the horizontal line is labeled "worst imaginable pain".
Time Frame: Day 30
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Iovera° Treatment | Sham Treatment
Number analyzed (Participants) | 112 | 56
percentage of participants | 67.9 | 48.2

7. Secondary Outcome: Change From Baseline in Total WOMAC Score at Day 60
Description: The WOMAC is a tri-dimensional, disease-specific, patient-reported outcome measure. It consists of 24 questions [each question is presented in a numerical rating scale format with possible values between 0= No (best) to 10= Extreme (worst)] with 5 questions regarding pain [possible subscale score 0 to 50], 2 questions regarding stiffness [possible subscale score 0 to 20] and 17 questions regarding function difficulty [possible subscale score 0 to 170]. The WOMAC total score was calculated by summing the 3 subscales for a total possible score of 0 to 240. A negative change from Baseline indicates improvement.
Time Frame: Baseline to Day 60
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Iovera° Treatment | Sham Treatment
Number analyzed (Participants) | 112 | 56
score on a scale | -70.50 (5.52) | -49.99 (7.81)

8. Secondary Outcome: VAS Responder Rate at Day 60
Description: VAS Responder Rate is defined as the percentage of participants with at least a 30% reduction in VAS at Day 60 compared to Baseline. VAS pain assessment is a measure of pain intensity. The scale is made up of a 10 cm (100 mm) horizontal line. The far left of the horizontal line is labeled "no pain" while the far right of the horizontal line is labeled "worst imaginable pain".
Time Frame: Day 60
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Iovera° Treatment | Sham Treatment
Number analyzed (Participants) | 112 | 56
percentage of participants | 65.2 | 55.4

9. Secondary Outcome: WOMAC Pain Score Responder Rate at Day 60
Description: WOMAC Pain Score Responder Rate is defined as the percentage of participants with at least a 30% reduction in the WOMAC pain score at Day 60 compared to Baseline. WOMAC is a tri-dimensional, disease-specific, patient-reported outcome measure. It consists of 24 questions [each question is presented in a numerical rating scale format with possible values between 0= No (best) to 10= Extreme (worst)] with the first 5 questions regarding pain [possible subscale score 0 to 50].
Time Frame: Day 60
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Iovera° Treatment | Sham Treatment
Number analyzed (Participants) | 112 | 56
percentage of participants | 64.3 | 48.2

ADVERSE EVENTS:
Time Frame: 6 Months
Description: Adverse Event (AE) data was collected over a 6 month period. Patients were followed until AE's were resolved.
Arm/Group | Iovera° Treatment | Sham Treatment
All-Cause Mortality (participants affected / at risk) | 1/121 | 0/59
Serious Adverse Events (participants affected / at risk) | 2/121 | 1/59
Other Adverse Events (participants affected / at risk) | 121/121 | 59/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Iovera° Treatment (N=121) | Sham Treatment (N=59)
Myocardial infarction (Cardiac disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Iovera° Treatment (N=121) | Sham Treatment (N=59)
Administration site bruise (Skin and subcutaneous tissue disorders) | 93 | 31
Administration site dysaesthesia (Skin and subcutaneous tissue disorders) | 25 | 11
Administration site pain (Skin and subcutaneous tissue disorders) | 26 | 11
Administration site paraesthesia (Skin and subcutaneous tissue disorders) | 17 | 2
Administration site scab (Skin and subcutaneous tissue disorders) | 6 | 3
Administration site swelling (Skin and subcutaneous tissue disorders) | 49 | 16
Application site discolouration (Skin and subcutaneous tissue disorders) | 1 | 0
Application site pruritus (Skin and subcutaneous tissue disorders) | 7 | 2
Application site hypoaesthesia (Skin and subcutaneous tissue disorders) | 63 | 32
Application site erythema (Skin and subcutaneous tissue disorders) | 50 | 24
Application site pain (Skin and subcutaneous tissue disorders) | 46 | 23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No